CLINICAL TRIAL: NCT03414541
Title: A Randomised, Double-Blind, Placebo-Controlled, Exploratory Phase IIa Study To Assess The Safety And Efficacy Of Orally Administered DS102 In Chronic Obstructive Pulmonary Disease Patients
Brief Title: Safety And Efficacy Study Of Orally Administered DS102 In Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afimmune (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DS102A-03
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants in this group will receive matching placebo capsules twice daily.
  Interventions: Other: Placebo
- 500mg DS102 (Experimental): Participants in this group will receive 500 mg DS102 capsules twice daily.
  Interventions: Drug: DS102
- 1000mg DS102 (Experimental): Participants in this group will receive 1000 mg DS102 capsules twice daily.
  Interventions: Drug: DS102

INTERVENTIONS:
Drug: DS102 — DS102
  Arms: 1000mg DS102; 500mg DS102
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this randomised, double-blind, placebo-controlled, parallel group study is to assess the safety and efficacy of orally administered DS102 capsules versus placebo in the treatment of adult patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) aged 40-75 years with stable COPD at the time of screening.
* Patients who are current or ex-smokers who have a smoking history of at least 10 pack years (Ten pack- years are defined as 20 cigarettes a Day for 10 years, or 10 cigarettes a Day for 20 years).
* Patients whose pre-study clinical laboratory findings do not interfere with their participation in the study, in the opinion of the Investigator.
* Patients who are able to communicate well with the Investigator, to understand and comply with the requirements of the study, and understand and sign the written informed consent.

Exclusion Criteria:

* Patients with a history of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* Patients with significant systemic or major illness other than pulmonary disease, including coronary artery disease, liver disease, cerebrovascular disease, renal insufficiency, serious psychiatric disease, respiratory or hypertensive disease, as well as diabetes and arthritis that, in the opinion of the Investigator, would preclude the patient from participating in and completing the study.
* Patients with known hypersensitivity to any ingredients of the study treatment.
* Patients, in the opinion of the Investigator, not suitable to participate in the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-09-24 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Change in induced sputum differential neutrophil count from baseline to Week 12 | 12 weeks
Number of Treatment Emergent Adverse Events (TEAEs) in each treatment group leading to treatment discontinuation. | 12 Weeks

SECONDARY OUTCOMES:
Change in induced sputum neutrophil differential count from baseline | 14 weeks
Change in St Georges Respiratory Questionnaire (SGRQ) from baseline | 14 weeks
  Questionnaire designed to measure impact of COPD on overall health, daily life and perceived well-being. Scores range from 0 -100 with higher scores indicating more limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Pavord, MA DM FRCP FERS FMedSci, Principal Investigator — University of Oxford, Oxford, UK
Locations (3):
- United Kingdom (3):
  - UK Site 2, Belfast
  - UK Site 3, London
  - UK Site 1, Manchester